CLINICAL TRIAL: NCT02319720
Title: A Randomized Study to Evaluate the Safety of Bone Marrow Aspirate Plus Cultured Bone Marrow Cells vs. Bone Marrow Aspirate Alone vs. Cultured Bone Marrow Cells Alone in the Treatment of Chronic Wounds.
Brief Title: Study to Evaluate Bone Marrow Cells in the Treatment of Chronic Wounds
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Dr. E.Badiavas (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Dr. E.Badiavas, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080299; 5R01AG027874 (NIH)
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Ulcer
MeSH Terms: conditions — Ulcer | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BMA/Cultured Bone Marrow Cells (Experimental): The subjects in this arm will have fresh bone marrow aspirate administered to the wound at the time the bone marrow is taken. Part of the aspirate will be cultured. Up to three applications of cultured cells will be applied to the wound following the bone marrow biopsy. A single treatment cycle will consist of one application of a freshly obtained bone marrow aspirate and up to three applications of cultured cells derived from that aspirate. If the wound has not healed, up to three additional treatment cycles may be performed. Each bone marrow biopsy will be followed by direct application of fresh bone marrow to the wound and up to three applications of cultured cells (prepared from the most recent bone marrow biopsy).
  Interventions: Biological: Bone Marrow Aspirate; Biological: Cultured Bone Marrow Cells; Procedure: Control
- Cultured Bone Marrow Cells (Experimental): In this group, the bone marrow aspirate will be sent to the laboratory to be grown in tissue culture. Once the cell cultures have matured (within 8 weeks) they will be checked for sterility and frozen until applied to the subject's wound. Up to three applications of cultured cells will be applied to the wound following the bone marrow biopsy. A single treatment cycle will consist of up to three applications of cultured cells derived from a single bone marrow aspiration. If the wound has not healed, up to three additional treatment cycles may be performed. Each bone marrow biopsy will be followed by up to three applications of cultured cells (prepared from the most recent bone marrow biopsy).
  Interventions: Biological: Cultured Bone Marrow Cells; Procedure: Control
- Bone Marrow Aspirate (Experimental): The subjects in this group will have fresh bone marrow aspirate administered to the wound at the time the bone marrow is taken. A single treatment cycle will consist of one application of a freshly obtained bone marrow aspirate. If the wound has not healed, up to three additional bone marrow biopsies may be performed. If the wound heals at any point during this protocol, no additional bone marrow biopsy procedures will be performed and no additional cells will be applied.
  Interventions: Biological: Bone Marrow Aspirate; Procedure: Control
- Control (Active Comparator): In this arm, subjects will receive currently approved treatments for their wound. These treatments will include debridement and dressing changes. Wound dressings allowed will include gauze, foam dressings, occlusive films, and non-stick pads. More advanced dressing materials such as Hydrocolloids, alginates, silver containing dressing and biomaterials can also be used. Compression will be utilized for lower extremity wounds.
  Interventions: Procedure: Control

INTERVENTIONS:
Biological: Bone Marrow Aspirate — Fresh bone marrow aspirate administered to the wound at the time the bone marrow is taken.
  Arms: BMA/Cultured Bone Marrow Cells; Bone Marrow Aspirate
Biological: Cultured Bone Marrow Cells — The bone marrow aspirate will be sent to the laboratory to be grown in tissue culture. Once the cell cultures have matured (within 8 weeks) they will be checked for sterility and frozen until applied to the subject's wound.
  Arms: BMA/Cultured Bone Marrow Cells; Cultured Bone Marrow Cells
Procedure: Control — The subjects in this group will receive currently approved treatments for their wound. These treatments will include debridement and dressing changes. Wound dressings allowed will include gauze, foam dressings, occlusive films, and non-stick pads. More advanced dressing materials such as Hydrocolloids, alginates, silver containing dressings, and biomaterials can also be used. Compression will be utilized for lower extremity wounds.
  Other Names: Standard of Care

SUMMARY:
Management of chronic wounds with:

1. Bone Marrow Aspirate Plus Cultured Cells Group
2. Cultured Cells Alone Group
3. Bone Marrow Aspirate Alone Group
4. Control Group

DETAILED DESCRIPTION:
Prior to randomization the subject will be screened for HIV, Hepatitis B and Hepatitis C. Women of child bearing age will be tested for pregnancy. As this is primarily a safety study, an electrocardiogram is done at the start of the study as a baseline in order to document any potential changes at a later date.

After the initial randomization visit the subject will return to have the wound examined once a week for 17 weeks after each treatment cycle begins or until the wound heals, whichever is earlier. Up to 4 treatment cycles will be allowed. As soon as the wound is completely healed, the subject will return once a month for 6 months to be certain the wound remains healed. The duration of the subject wound participation in the study is expected to be a maximum of 18 months following the start of study treatment.

The subjects in this study will be randomized into one of four arms. Three groups will receive bone marrow cells and one will not receive bone marrow cells (control group).

1. Bone Marrow Aspirate (BMA) Plus Cultured Cells Group:

   The subjects in this arm of the study will have fresh bone marrow aspirate administered to the wound at the time the bone marrow is taken. Part of the aspirate will be cultured. Once the cell cultures have matured (within 8 weeks) they will be checked for sterility, and frozen until applied to the wound. Up to three applications of cultured cells will be applied to the wound following the bone marrow biopsy. A single treatment cycle will consist of one application of a freshly obtained bone marrow aspirate and up to three applications of cultured cells derived from that aspirate. If the wound has not healed, up to three additional treatment cycles may be performed. Each bone marrow biopsy will be followed by direct application of fresh bone marrow to the wound and up to three applications of cultured cells (prepared from the most recent bone marrow biopsy). If the wound heals at any point during this protocol, no additional bone marrow biopsy procedures will be performed and no additional cells will be applied.
2. Cultured Cells Alone Group:

   In this group, the bone marrow aspirate will be sent to the laboratory to be grown in tissue culture. Once the cell cultures have matured (within 8 weeks) they will be checked for sterility and frozen until applied to the subject wound. Up to three applications of cultured cells will be applied to the wound following the bone marrow biopsy. A single treatment cycle will consist of up to three applications of cultured cells derived from a single bone marrow aspiration. If the wound has not healed, up to three additional treatment cycles may be performed. Each bone marrow biopsy will be followed by up to three applications of cultured cells (prepared from the most recent bone marrow biopsy). If the wound should heal at any point during this protocol, no additional bone marrow biopsy procedures will be performed and no additional cells will be applied.
3. Bone Marrow Aspirate Alone Group:

   The subjects in this group will have fresh bone marrow aspirate administered to the wound at the time the bone marrow is taken. A single treatment cycle will consist of one application of a freshly obtained bone marrow aspirate. If the wound has not healed, up to three additional bone marrow biopsies may be performed. If the wound heals at any point during this protocol, no additional bone marrow biopsy procedures will be performed and no additional cells will be applied.
4. Control Group

The subjects in this group will receive currently approved treatments for their wound. These treatments will include debridement and dressing changes. Wound dressings allowed will include gauze, foam dressings, occlusive films, and non-stick pads. More advanced dressing materials such as hydrocolloids, alginates, silver containing dressing, and biomaterials can also be used. Compression will be utilized for lower extremity wounds.

VISIT SCHEDULING; Regardless of the group the subject is assigned to, he/she will be asked to return weekly for Standard Of Care (SOC) and wound evaluation. Subjects that miss more than 4 consecutive weekly visits and are not receiving SOC elsewhere, may be removed from the study. After this (or after wound closure if this occurs earlier) the subject will return once a month for 6 months for evaluation.

Follow-up study visits will be arranged at 1 to 4 week intervals based on clinical evaluations and scheduling restrictions until the wound heals.

Once the wound is determined to have healed, the subject will be asked to return monthly for 6 months to be certain the wound remains healed.

Subjects with non-healing wounds will be monitored for 6 months following the last administration of bone marrow cells.

Lower extremity wounds will be covered with a compression bandage. If a wound is not located on a lower extremity, it will be covered by a nonstick pad, an adsorbent pad, a gauze wrap and, optionally, a light compression bandage.

Subjects with diabetic wounds will be asked to submit a record of blood sugar monitoring. The blood levels of Hemoglobin A1c will also be monitored at three-month intervals if this is not already being done routinely. If the Hemoglobin A1c levels are above 10%, the physician who is managing the subject diabetes will be contacted to discuss any changes in medication to control the subject diabetes.

All study examinations will include observation of healing, wound tracing measurements and photography of the wound.

All subjects will have a skin biopsy taken at the time of healing or at the week 17 end of treatment cycle visit. Tissues derived from debridement procedures will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age or older with chronic wounds
2. Wound present for at least one year
3. Subjects must understand and give written informed consent.
4. Subjects must agree to have biopsies performed as per protocol
5. Subjects must be accessible for weekly wound treatment and assessment visits
6. Patients with chronic osteomyelitis will be eligible. They must however be afebrile, and have completed a 6-week course of intravenous and/or oral antibiotics. The use of chronic suppressive antibiotics will be allowed.

Exclusion Criteria:

1. Have evidence of active infection at the wound site
2. Evidence of active malignancy in ulcer
3. Have any requirement for the use of systemic steroids or immunosuppressive agents
4. Be a pregnant female or nursing mother
5. Subjects who are known or found to be HIV positive
6. Evidence of dry/wet gangrene
7. History of alcohol or substance abuse within the past 18 months
8. Patients with severe medical conditions

   1. Malignancy (other than non melanoma skin cancer) not in remission or in remission less than 5 years
   2. Life expectancy less than two years
   3. Severe cardiopulmonary disease restricting ambulation to the clinical facility
9. Severe arterial or vascular disease requiring or best treated by amputation
10. Untreated osteomyelitis affecting the ulcer area or osteomyelitis affecting the ulcer area not receiving aggressive treatment
11. History of poor compliance, unreliability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-07; Primary Completion 2013-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety Bone Marrow Fresh Cells directly to wounds (Number of adverse events) | 12 months
  Number of adverse events reported
Safety Bone Marrow Cultured Cells directly to wounds (Number of adverse events) | 12 months
  Number of adverse events reported
Safety Bone Marrow Cultured Cells and Bone Marrow fresh cells directly to wounds (Number of adverse events) | 12 months
  Number of adverse events reported

SECONDARY OUTCOMES:
Efficacy Bone Marrow Fresh Cells in wounds (Healing rate) | 12 months
  Healing rate of wounds at end of participation
Efficacy Bone Marrow Cultured Cells in wounds (Healing rate) | 12 months
  Healing rate of wounds at end of participation
Efficacy Bone Marrow Cultured Cells and Bone Marrow Fresh Cells in wounds (Healing rate) | 12 months
  Healing rate of wounds at end of participation

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos V Badiavas, MD, PhD, Principal Investigator — University of Miami